CLINICAL TRIAL: NCT03495804
Title: Evaluation of the Performance of Two Neutral Oral Contrast Agents in CT Enterography (CTE)
Brief Title: Evaluation of the Performance of Two Neutral Oral Contrast Agents in CT Enterography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018SDU-QILU-01
Record Dates: First submitted 2018-01-13; First posted 2018-04-12 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: CTE
Keywords: CT enterography; oral contrast agent
MeSH Terms: interventions — Polyethylene Glycols; Mannitol

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to group A or B. Participants of group A are given isotonic mannitol as oral contrast agent, while participants of group B are given isotonic polyethylene glycol as oral contrast agent.
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mannitol (Active Comparator): Participants are given a minimum of 1500 mL of a preparation of mannitol as oral contrast agent over an hour prior to the examination.
  Interventions: Drug: mannitol
- polyethylene glycol (Experimental): Participants are given a minimum of 1500 mL of a preparation of polyethylene glycol as oral contrast agent over an hour prior to the examination.
  Interventions: Drug: polyethylene glycol

INTERVENTIONS:
Drug: polyethylene glycol — Experimental group was given polyethylene glycol as oral contrast agent.
  Arms: polyethylene glycol
Drug: mannitol — Active comparator group was given mannitol as oral contrast agent.
  Arms: mannitol

SUMMARY:
CT enterography has become an important tool in the evaluation of small bowel diseases, especially in patients with inflammatory bowel diseases. There are several shortcomings of commonly used isotonic mannitol as an oral contrast agent, such as incident adverse reactions and gases in the gut. However, polyethylene glycol can avoid these drawbacks with a good performance in some pilot experiments.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 to 75
* patients undergoing CT enterography

Exclusion Criteria:

* patients with a history of colorectal surgery
* patients with severe colonic stricture or obstructing tumor
* patients with significant gastroparesis or gastric outlet obstruction
* patients with known or suspected bowel obstruction or perforation
* patients with severe chronic renal failure (creatinine clearance<30 ml/min)
* patients with uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* patients with severe inflammatory bowel disease or megacolon
* patients with documented allergy to intravascular contrast agent
* patients with dehydration
* patients with pregnancy or lactation
* patients hemodynamically unstable
* patients with dysphagia
* patients with severe constipation.
* patients unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Performance of two neutral oral contrast agents in CT enterography. | 12 months
  The assessment system includes six parts.
  1. Whether the contrast reached the caecum is evaluate and recorded as 'yes' or 'no'.
  2. The overall presence of inhomogeneous contrast is evaluated and recorded as 'yes' or 'no'.
  3. The maximum dimension of a single loop in each quadrant was recorded.
  4. The scale of loops of small bowel distended ≥2 cm are evaluated and recorded as '0-25%', '26-50%', '51-75%' and '76-100%'.
  5. The wall visibility and visualization of the small-bowel mucosal are scored on a scale ranging from 1 to 4, in which a higher score represents a better outcome.
  6. Overall quality is assessed subjectively by the radiologist and scored on a scale ranging from 1 to 4, in which a higher score represents a better outcome.

SECONDARY OUTCOMES:
Side effects of the two oral contrast agents. | 12 months
  The degree of nausea, emesis, diarrhea, abdominal distension and cramp following ingestion are scored on a scale ranging from 0 to 10, in which a higher score represents a higher level of these targets.
The flavor, volume and participants' willing for the second use of the two oral contrast agents in CT enterography. | 12 months
  The flavor, volume and participants' willing for the second use are scored on a scale ranging from 0 to 10, in which a higher score represents a better outcome.
Dizziness and debilitation of patients. | 12 months
  The presence of dizziness and debilitation are recorded as 'yes' or 'no'.
Temperature of patients. | 12 months
  The temperature of patients are recorded in degree centigrade.
Blood pressure of patients. | 12 months
  The blood pressure of patients are recorded in millimeter of mercury.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China